CLINICAL TRIAL: NCT06613568
Title: Prospective, Non-Randomized, Multicenter, Open-Label Study Evaluating the Use of the Moda-flx Hemodialysis System™ Under Professional Care and At Home by Participants With End Stage Kidney Disease (ESKD) Who Are on Stable Dialysis Regimens
Brief Title: Moda-flx Hemodialysis System™ Under Professional Care Settings by Trained Individuals and At Home by Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diality Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIA-HHD-001
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: End Stage Kidney Disease
Keywords: Renal Disease; Hemodialysis Complication; Kidney Diseases; Dialysis; Renal Dialysis; Hemodialysis, Home; Renal Insufficiency; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Professional Care and At Home (Experimental): Participants will receive dialysis therapy using the Moda-Flx Hemodialysis System™ in a Professional Care setting and At Home setting
  Interventions: Device: Moda-flx Hemodialysis System™

INTERVENTIONS:
Device: Moda-flx Hemodialysis System™ — The Moda-flx Hemodialysis System™ is a portable hemodialysis system

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Moda-flx Hemodialysis System™ when used Under Professional Care Settings by trained individuals and At Home by trained Participants and Care Partners

ELIGIBILITY:
Inclusion Criteria:

* Are between 18 and 80 years of age and Care Partner is at least 18 years of age at the time of signing consent.
* Have a diagnosis of end stage kidney disease (ESKD) adequately treated by maintenance dialysis (defined as achieving a spKt/V ≥ 1.2 OR stdKt/V ≥ 2.1) and be deemed stable by their treating nephrologist prior to the end of the Screening Period
* Have a well-functioning and stable vascular access (tunneled central venous catheter arteriovenous fistula, or graft) that allows a blood flow of at least 300 ml/min prior to the end of Screening
* Can successfully complete a Skills and Comprehension Assessment with a Care Partner prior to the completion of the Training Period.

Exclusion Criteria:

* Hgb level of < 9 g/dL at Screening
* Symptomatic intradialytic hypotension requiring medical intervention (ultrafiltration turned off, bolus of fluid) in at least two treatments during the Run-In period defined as:

  1. Persistent pre-dialysis sitting SBP < 100 mmHg despite medical therapy,
  2. Nadir intradialytic Systolic Blood Pressure (SBP) < 90 mmHg, if Subject's pre-HD SBP < 160 mmHg
  3. Nadir intradialytic SBP < 100 mmHg if Subject's pre-HD SBP ≥ 160 mmHg
* Documented history of non-adherence to dialysis therapy that would prevent successful completion of the study
* Participant had an average ultrafiltration rate > 13 mL/kg/hour during the last 2 weeks prior to Screening, per medical records.
* Had a significant cardiovascular adverse event within the last 90 days prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Weekly Standardized Dialysis Adequacy | Up to 10 weeks per period
  Standardized weekly (stdKt/V) values as measured once every week during the Professional Care and At Home treatment settings
Adverse Event (AE) Rate | Up to 10 weeks per period
  The adverse event (AE) rate: defined as the number of Study Emergent AEs per 100 dialysis treatments occurring in the At Home period of the study, compared with those occurring during the Professional Care period.

SECONDARY OUTCOMES:
Goal Ultrafiltration Volume | Up to 10 weeks per period
  Compliance with fluid removal goals that are defined as:
  Ultrafiltration (net fluid removal), such that the recorded value from the Moda-flx Hemodialysis System™ is within ± 100 mL/h or ± 250 mL (whichever is less) of set point during the treatment, based on the UF prescription.
Study Emergent Pre-Specified Adverse Events | Up to 10 weeks per period
  Study Emergent Pre-Specified Adverse Eventss, categorized by study period (Professional Care and At Home) severity, device relationship and procedure relationship. Study-emergent Pre-Specified AEs are those AEs with an onset on or after the date of first treatment during the Run-In Period, which will be comprised of any of the following:
  1. A composite of:
  * Serious Adverse Event
  * Allergic Reaction
  * Blood Loss
  * Hemolytic Reaction
  * Infection
  * Intradialytic Event
  * Vascular Access Complication
  * Pyrogenic Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Silva, MD, Study Director — Diality Inc.
Locations (4):
- United States (4):
  - North America Research Institute, San Dimas, California
  - Nephrology Associates of Knoxville, Knoxville, Tennessee
  - aQua Research Institute, LLC, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No